CLINICAL TRIAL: NCT03504657
Title: Drug-coated Balloon Angioplasty for Patients With Symptomatic Vertebral Artery Stenosis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Zhengzhou University (Other)
Responsible Party: Principal Investigator, Chuanjie Wu, MD, The First Affiliated Hospital of Zhengzhou University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FAHZU-2018-006
Record Dates: First submitted 2018-04-12; First posted 2018-04-20 (Actual); Last update posted 2018-05-04 (Actual); Status verified 2018-05

CONDITIONS: Vertebral Artery Stenosis
Keywords: Vertebral Artery Stenosis; Drug-coated balloon angioplasty; Stenting
MeSH Terms: conditions — Vertebrobasilar Insufficiency

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Drug-coated balloon angioplasty (Experimental)
  Interventions: Device: Drug-coated balloon angioplasty
- stenting angioplasty (Active Comparator)
  Interventions: Device: stenting angioplasty

INTERVENTIONS:
Device: Drug-coated balloon angioplasty — Angioplasty with a drug-coated angioplasty
  Arms: Drug-coated balloon angioplasty
Device: stenting angioplasty — Angioplasty with a stenting
  Arms: stenting angioplasty

SUMMARY:
Posterior circulation stroke accounts for 20% of ischemic stroke. A quarter occurs in patients with stenosis in the vertebral and/or basilar arteries. Vertebral artery stenosis can be treated with stenting. However, in-stent restenosis rate have been reported as high as more than 30%, which may reduce the effect of stent therapy. Drug-coated balloon has shown good results in controlling neointimal hyperplasia in the femoral and popliteal arteries.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Patients presenting with posterior circulation transient ischemic attack or nondisabling stroke in the previous 6 months
* Vertebral artery origin stenosis resulting from presumed atheromatous disease with stenosis ≥50%
* Lesion length of the stenosis >5mm.
* Angioplasty can be performed within two weeks after randomization
* Female subjects of childbearing potential have a negative pregnancy test.
* Signed informed consent prior to entering study

Exclusion Criteria:

* Potential cause of TIA or minor stroke other than stenosis in a vertebral artery (e.g. atrial fibrillation)
* Life expectancy shorter than 2 years
* Vertebral artery stenosis caused by dissection
* Vertebral stenting felt to be technically impracticable
* Previous stenting in randomized artery
* Pre-morbid modified Rankin scale score of greater than 3
* Currently participating or previously participated in any investigational drug or device study within 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2018-05-03 (Actual); Primary Completion 2019-05-01 (Estimated); Study Completion 2020-04-30 (Estimated)

PRIMARY OUTCOMES:
Restenosis | 12 months

SECONDARY OUTCOMES:
The composite of vascular death, myocardial infarction, or any stroke | within 30 days after the start of treatment
The composite of vascular death, myocardial infarction, or any stroke | within 12 months after the start of treatment
Death resulting from any cause | 12 months
Stroke in the supply territory of the symptomatic vertebral artery | 12 months

OTHER OUTCOMES:
Serious adverse events | 30 days

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Nanyang City Center Hospital, Nanyang